CLINICAL TRIAL: NCT04607863
Title: Foot Posture Index Pronated, Hallux Limitus Connection and Chronic Low Back Pain Gait Parametrers With Optogait Sensor
Brief Title: Foot Posture Index, Hallux Limitus in Patients With Chronic Low Back Pain. Gait With Optogait Sensor
Status: Completed | Type: Observational
Sponsor: University of Seville (Other)
Responsible Party: Principal Investigator, Aurora Castro Mendez, Aurora Castro-Méndez, University of Seville
Other Study IDs: 23/11
Record Dates: First submitted 2020-10-23; First posted 2020-10-29 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2020-01

CONDITIONS: Hallux Limitus; Movement, Abnormal; Back Pain Lower Back Chronic
Keywords: foot; hallux; limitus; back
MeSH Terms: conditions — Hallux Limitus; Dyskinesias

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Low back pain: Patients with low back pain
  Interventions: Diagnostic Test: Case control
- No low back pain: No low back pain patients
  Interventions: Diagnostic Test: Case control

INTERVENTIONS:
Diagnostic Test: Case control — Is a case-control research

SUMMARY:
Foot disorders have been recognized as being linked to chronic low back pain

DETAILED DESCRIPTION:
Foot disorders have been recognized as being linked to chronic low back pain (CLBP), To improve knowledge of the relationship between the limitation of the movement range of hallux (HROML) is important about it can affect the back biomechanical . The aim of this research is to investigate if the HROML may appear as a risk factor of CLBP

HROML affect the foot position, and consecuently may induce to alter as compensatory mechanism the normal biomechanical of the leg, hip and back.

ELIGIBILITY:
Inclusion Criteria: males and females between 18 to 65 years old Hallux limitus in one or two feet -

Exclusion Criteria:

serious illness, current participation in another research study pregnancy previus foot or back surgery

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Males and females between 18 and 65 years old
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-01-23 (Actual); Primary Completion 2020-11-02 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Hallux dorsal movement range degrees | A day, the inclusion day in the study
  Goniometer to examinate the range of hallux dorsal movement

SECONDARY OUTCOMES:
Low back pain | a day, the inclusion day in the study
  questionnary oswestry disability index

CONTACTS AND LOCATIONS:
Locations (1):
- Aurora Castro Mendez, Seville, Spain

IPD SHARING:
Plan to Share IPD: No